CLINICAL TRIAL: NCT06885385
Title: An Open-label, Multicenter, Phase 2 Clinical Study Evaluating the Safety and Efficacy of JS207 With or Without JS015 in Combination With Chemotherapy (XELOX) as First-line (1L) Treatment in Patients With MSS/pMMR Advanced Colorectal Cance
Brief Title: A Phase 2 Study Evaluating the Safety and Efficacy of JS207 With or Without JS015 in Combination With Chemotherapy in Patients With Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS207-007-II-CRC
Record Dates: First submitted 2025-03-09; First posted 2025-03-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS207 (Experimental)
  Interventions: Biological: JS207; Biological: JS015; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: JS207 — JS207 will be administered every 3 weeks for a treatment cycle of 21 days
Biological: JS015 — JS015 will be administered every 3 weeks for a treatment cycle of 21 days
Drug: Capecitabine — Capecitabine of 1000mg/m2 will be administered orally twice daily from day 1 to 14 every 21 day cycle
Drug: Oxaliplatin — Oxaliplatin of 130mg/m2 will be administered intravenously (IV) on day 1 every 21 day cycle

SUMMARY:
This study is an open label, multicenter Phase II clinical trial aimed at evaluating the safety and efficacy of JS207 with or without JS015 in combination with chemotherapy (XELOX) as a first-line treatment for advanced colorectal cancer with MSS/pMMR. The study was divided into two cohorts: Cohort 1 was JS207 combined with XELOX, and Cohort 2 was JS207 combined with JS015 and XELOX.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 75 (inclusive) at the time of signing the consent form, both male and female
2. Colorectal adenocarcinoma or rectal adenocarcinoma with histological or cytological Qualification, according to the 8th edition of the AJCC colorectal cancer TNM staging stage IV, MSS/pMMR (a qualified report of MSS or pMMR detected by a local laboratory must be provided), and no previous systemic anti-tumor therapy for advanced disease; for patients who have received neoadjuvant or adjuvant systemic therapy, the last treatment to relapse or progression takes more than 12 months
3. ECOG score is 0 or 1
4. Estimated survival ≥ 12 weeks
5. According to the RECIST v1.1 evaluation standard, there is at least one measurable lesion
6. Good organ function
7. Female or male subjects with fertility must agree to have no family planning during the study period and voluntarily use effective contraception with significant others within 6 months after the end of the last medication. Female subjects with fertility (WOCBP) must have a negative serum pregnancy test within 7 days before the first medication and be non-lactating (see section 10.3 for specific contraceptive measures and WOCBP definitions)
8. The patient participated voluntarily, gave full informed consent, signed a written ICF, and had good compliance

Exclusion Criteria:

1. Previously received PD-1 or programmed cell death ligand 1 (PD-L1) inhibitor therapy; or previously received DKK1 inhibitor therapy (only for cohort 2 subjects)
2. Received the following medications or treatments before the first dose Within 28 days before the first dose, major surgery and radiotherapy (palliative radiotherapy for local bone/brain lesions, allowed to be completed within 14 days before the first dose) were performed. Within 7 days before the start of the study, coarse needle aspiration biopsy or other minor surgery was performed, excluding the placement of vascular infusion devices.

   Within 14 days before the first medication, antiplatelet therapy such as aspirin (≥ 325 mg/day), clopidogrel (≥ 75 mg/day), or anticoagulant therapy for therapeutic purposes have been used.

   Patients who have received systematic treatment with corticosteroids (> 10 mg prednisone or equivalent dose per day) or other immunosuppressants for more than 1 week before the first dose are allowed to use inhaled or topical steroids or ≤ 10 mg/day systemic prednisone and equivalent doses of similar drugs for treatment.

   D) Have received any live vaccine or attenuated live vaccine within 28 days before the first dose, or expect to receive live vaccine or attenuated live vaccine during the study period (limited to patients in combination therapy studies);
3. The toxicity of previous anti-tumor treatment has not been restored to the level specified in CTCAE v5.0 or the level specified in the inclusion/exclusion criteria, except for the following cases: the relevant toxicity that has been judged by the investigator to be well controlled and does not affect the safety and compliance of the patient with the study drug can be screened after qualification with the sponsor
4. Digestive tract perforation, fistula, abdominal abscess, and digestive system ulcerative diseases or a history thereof within 6 months prior to the first medication (the investigator may consider inclusion if the ulcer condition is stable)
5. There are pleural effusion, abdominal effusion or pericardial effusion with clinical symptoms that require repeated treatment (puncture or drainage, etc.)
6. History of interstitial lung disease or previous history of non-infectious pneumonia treated with corticosteroids, or evidence of active pneumonia on screening imaging
7. Severe, unhealed or open wounds, active ulcers, or untreated fractures (excluding old fractures evaluated by researchers as not requiring clinical intervention)
8. Evidence of obvious bleeding tendency or severe coagulation dysfunction,Have a history of gastrointestinal bleeding within the 6 months prior to enrollment, or have a clear tendency towards gastrointestinal bleeding (including severe esophageal-gastric varices with bleeding risk, locally active gastrointestinal ulcer lesions, and persistent positive fecal occult blood),Clinically significant hemoptysis or tumor bleeding for any reason within 28 days before the first medication.Screening period imaging shows that the tumor surrounds important blood vessels or has obvious necrosis and cavities, and the researchers believe that it may cause bleeding risks
9. Presence of poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure > 100 mmHg), or a history of hypertensive crisis or hypertensive encephalopathy
10. Severe cardiovascular and cerebrovascular diseases, including but not limited to: myocardial infarction, severe/unstable angina pectoris, congestive heart failure (New York Heart Association [NYHA] heart function classification ≥ 2), clinically significant supraventricular or ventricular arrhythmia requiring drug intervention, aortic aneurysm requiring surgical repair, any arterial thrombosis/embolism events, grade 3 or above (CTCAE v5.0) venous thrombosis/embolism events, transient cerebral ischemic attack, cerebrovascular accident; left ventricular ejection fraction (LVEF) < 50% in cardiac ultrasound examination. The corrected QT interval (QTc) is > 480 ms (calculated using the Fridericia method. If the QTc is abnormal, it can be detected three times continuously every 2 minutes and the average value is taken)
11. There is active Central Nervous System metastasis. If the patient has received radiotherapy or surgery in the past, the imaging examination within 4 weeks before the first medication shows that the brain metastasis is stable and there is no aggravation or new neurological symptoms. Hormonal therapy has been stopped two weeks before the first medication, and screening is allowed; for the presence of meningeal metastasis and brainstem metastasis, screening is not allowed regardless of treatment
12. Severe infection (CTCAE v5.0 > 2) occurred within 28 days before the first study administration, such as severe pneumonia, bacteremia, and comorbidities requiring hospitalization; or active infection requiring systemic anti-infective treatment or fever of unknown cause > 38.5 ℃ occurred within 2 weeks before the first study administration (according to the investigator's judgment, subjects with fever caused by tumors can be enrolled);
13. Active tuberculosis, hepatitis B (hepatitis B surface antigen [HBsAg] positive and HBV DNA higher than 1000 copies/ml or 200 IU/ml), hepatitis C (hepatitis C antibody [HCVAb] positive and HCV RNA higher than the lower limit of the research center)
14. Have a history of immunodeficiency diseases, including a positive test for human immunodeficiency virus (HIV), or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
15. Active autoimmune diseases that require systemic treatment (e.g. corticosteroids or immunosuppressive drugs) within 2 years before the first medication, including but not limited to: systemic systemic lupus erythematosus, multiple sclerosis, rheumatoid arthritis, inflammatory bowel disease, vasculitis, etc. However, thyroid, adrenal or pituitary gland dysfunction that can be controlled only with hormone replacement therapy, type 1 diabetes, psoriasis or vitiligo that do not require systemic treatment, childhood asthma/allergies that have been cured are allowed to be screened
16. Have a history of another primary malignant tumor, except for malignant tumors (such as basal cell carcinoma and squamous cell carcinoma of the skin that have received potential curative treatment) that have received radical treatment before the first dose of the study intervention and have no known active disease (more than 5 years) and low potential recurrence risk
17. Patients who have other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study, affect treatment adherence, or interfere with the study results, and are judged by the investigator to be unsuitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity （DLT) | 2 Years
  Incidence and severity of DLT
Adverse event（AE） | 2 Years
  Adverse events (AE), Abnormal changes in laboratory and other tests with clinical significance
RP3D | 2 Years
  Recommended dose for phase II trial
Objective response rate (ORR) based on Response Evaluation Criteria In Solid Tumors 1.1 (RECIST1.1) | 2 years
  Defined as the proportion of subjects who achieved partial response (PR) or complete response (CR)

SECONDARY OUTCOMES:
Progression free survival(PFS) | 2 years
  The time from first dose to Disease progression or death
Overall survival (OS) | 2 years
  The time from first dose to death from any cause
Immunogenicity | 2 years
  Incidence of Anti-Drug Antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai Oriental Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No